CLINICAL TRIAL: NCT05080192
Title: Cardiovascular, Pulmonary, and Integrative Functional Phenotypes in COVID-19 - Effect of Fenofibrate
Brief Title: Cardiovascular, Pulmonary, and Integrative Functional Phenotypes in COVID-19 Survivors - Effect of Fenofibrate
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 844349
Record Dates: First submitted 2021-08-17; First posted 2021-10-15 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Fenofibrate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, urine, breath condensate, buffy coat, endothelial cells and RNA will be collected from study subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fenofibrate recipients: Approximately 20 subjects who were randomized to the Fenofibrate arm in the FERMIN trial. This drug was administered for 10 days post-randomization.
  Interventions: Drug: Fenofibrate
- Placebo recipients: Approximately 20 subjects who were randomized to the placebo arm in the FERMIN trial. This drug was administered for 10 days post-randomization.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenofibrate — 145 mg/d of Tricor (administered as part of the parent FERMIN trial) for 10 days, or renal corrected dose equivalent (depending on renal function)
  Other Names: Tricor
  Groups: Fenofibrate recipients
Drug: Placebo — Matching placebo (once/day) for 10 days
  Groups: Placebo recipients

SUMMARY:
The International multicenter FEnofibRate as a Metabolic INtervention for COVID-19 (FERMIN) trial is being executed. The trial is testing a short intervention (10 days of fenofibrate therapy) on 30-day outcomes in COVID-19. The overarching goal of this sub-study is to explore the impact of fenofibrate on key longer term phenotypes of vascular, cardiac and pulmonary health, integrated cardiopulmonary function, persistent/chronic symptoms and quality of life.

DETAILED DESCRIPTION:
The International multicenter FEnofibRate as a Metabolic INtervention for COVID-19 (FERMIN) trial is being executed. The aim of this trial is to assess the impact of fenofibrate (administered for 10 days) to improve clinical outcomes in patients with COVID-19, assessed at 30 days. However, given the accumulating evidence of chronic / long term sequelae of COVID-19, it is important to assess the long-term impact of this intervention in this patient population. The overarching goal of this substudy is to assess the impact of fenofibrate on key intermediate phenotypes of vascular, cardiac and pulmonary health. We also aim to address the impact of fenofibrate therapy (administered during the acute COVID-19 episode as part of the parent FERMIN trial) on long-term integrated cardiopulmonary function, persistent/chronic symptoms and quality of life. We will accomplish this via enrollment of previous FERMIN participants from the University of Pennsylvania, in an phenotyping study designed to assess vascular, cardiac and pulmonary status several months after the index episode of COVID-19. We will perform these assessments ~6 months after initial randomization, among 40 FERMIN trial participants enrolled at the University of Pennsylvania.

ELIGIBILITY:
Inclusion Criteria:

• Having been eligible, enrolled and randomized in the parent FERMIN trial, completing all study procedures up to the 30-day time point (as specified in the parent protocol).

Exclusion Criteria

* Prisoners/incarcerated individuals;
* Pregnancy (potentially eligible patients of reproductive age will undergo a pregnancy test). This exclusion is due to the fact that pregnancy may confound the various cardiopulmonary phenotypes assessed in this study
* Inability to provide informed consent.
* History of cardiovascular disease (defined as heart failure, myocardial infarction, coronary revascularization, serious arrhythmia, stroke, or peripheral artery disease), glomerular disease or polycystic kidney disease prior to the index COVID-19 episode.
* Estimated glomerular filtration rate <30 mL/min/1.73m2 prior to the index COVID-19 episode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be screened from our FERMIN trial population. Participants will be approached by a member of the study team for participation. Participants will undergo a comprehensive assessment of key phenotypes (6±3 months after the index COVID-19 episode).
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fenofibrate Recipients: Participants who were randomized to the Fenofibrate arm in the FERMIN trial. This drug was administered for 10 days post-randomization.
  Fenofibrate: 145 mg/d of Tricor (administered as part of the parent FERMIN trial) for 10 days, or renal corrected dose equivalent (depending on renal function)
- Placebo Recipients: Participants who were randomized to the placebo arm in the FERMIN trial. This drug was administered for 10 days post-randomization.
  Placebo: Matching placebo (once/day) for 10 days
Period: Overall Study
Arm/Group | Fenofibrate Recipients | Placebo Recipients
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fenofibrate Recipients | Placebo Recipients | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.29 (10.64) | 40.2 (5.93) | 48.42 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Flow Mediated Dilation of the Brachial Artery
Description: Flow Mediated dilation of the brachial artery measured with ultrasound. This is a metric of endothelial function
Time Frame: At baseline visit
Population: The data for 1 fenofibrate recipient were omitted from analysis due to poor quality. 1 fenofibrate recipient did not undergo the test.
Measure: Median (Inter-Quartile Range); unit: % of brachial artery dilation
Arm/Group | Fenofibrate Recipients | Placebo Recipients
Number analyzed (Participants) | 5 | 5
% of brachial artery dilation | 6.1 [5.6 to 8.5] | 6.2 [5.0 to 10.6]

2. Primary Outcome: Arterial Wave Reflection Magnitude
Description: Arterial wave reflection magnitude measured with high fidelity arterial tonometry and wave separation analysis
Time Frame: At baseline visit
Population: The data for 1 fenofibrate recipient were omitted from analysis due to poor quality. 1 placebo recipient did not undergo the test.
Measure: Median (Inter-Quartile Range); unit: % of forward wave amplitude
Arm/Group | Fenofibrate Recipients | Placebo Recipients
Number analyzed (Participants) | 6 | 4
% of forward wave amplitude | 43.7 [37.9 to 51.8] | 42.9 [32.8 to 47.2]

3. Primary Outcome: Large Artery Stiffness
Description: Carotid-femoral pulse wave velocity measured with arterial tonometry
Time Frame: At baseline visit
Population: The data for 1 fenofibrate recipient was omitted due to poor quality. The data for 1 placebo recipient was not collected due to technical difficulty.
Measure: Median (Inter-Quartile Range); unit: m/s
Arm/Group | Fenofibrate Recipients | Placebo Recipients
Number analyzed (Participants) | 6 | 4
m/s | 5.8 [5.5 to 6.6] | 7 [5.4 to 8.4]

4. Primary Outcome: Myocardial Function
Description: Peak longitudinal strain assessed with echocardiography. Longitudinal strain was measured as the shortening of the LV cavity longitudinal dimension (mitral annulus plane to apex) in apical echocardiographic views, expressed as the percent change relative to the end-diastolic length, where shortening is expressed as a negative change.
Time Frame: At baseline visit
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: % change in length
Arm/Group | Fenofibrate Recipients | Placebo Recipients
Number analyzed (Participants) | 6 | 4
% change in length | -14.1 [-14.6 to -11.4] | -17.9 [-18.8 to -17.4]

5. Primary Outcome: Diffusion Capacity of Lungs for Carbon Monoxide (DLCO)
Description: Diffusion capacity of lungs for carbon monoxide (DLCO) measured during pulmonary function testing
Time Frame: At baseline visit
Population: The data for 2 participants (1 fenofibrate recipient and 1 placebo recipient) were omitted from analysis due to poor quality.
Measure: Median (Inter-Quartile Range); unit: mL/min/mmHg
Arm/Group | Fenofibrate Recipients | Placebo Recipients
Number analyzed (Participants) | 6 | 4
mL/min/mmHg | 23.3 [14.9 to 32.8] | 24 [19.5 to 32.1]

6. Primary Outcome: Aerobic Capacity
Description: Subjects will perform a maximal-effort peak oxygen consumption test using a supine bicycle exercise test with expired gas analysis.
Time Frame: At baseline visit
Population: 5 participants (2 fenofibrate recipients and 3 placebo recipients) did not undergo the test.
Measure: Median (Inter-Quartile Range); unit: mL/min/kg
Arm/Group | Fenofibrate Recipients | Placebo Recipients
Number analyzed (Participants) | 5 | 2
mL/min/kg | 12.1 [8.4 to 16.5] | 11.8 [10.0 to 13.6]

7. Primary Outcome: Self-reported Quality of Life Via Survey
Description: Quality of life measured with the Kansas City Cardiomyopathy questionnaire (KCCQ). The overall summary score from the KCCQ ranges from 0-100, where higher scores indicate a better quality of life.
Time Frame: At baseline visit
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fenofibrate Recipients | Placebo Recipients
Number analyzed (Participants) | 7 | 5
score on a scale | 75.7 [22.1 to 87.8] | 79.7 [74.5 to 81.5]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant starting on their baseline visit, during 24-hour ambulatory blood pressure monitoring, and at bike test, up to 3 days.
Description: Total number at risk is the total number of participants enrolled.
Arm/Group | Fenofibrate Recipients | Placebo Recipients
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 1/7 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenofibrate Recipients (N=7) | Placebo Recipients (N=5)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arm numbness (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The sample size of the study is too small (N=12) and there is not sufficient power to infer differences between the groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT05080192/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT05080192/ICF_001.pdf